CLINICAL TRIAL: NCT05353569
Title: Otitis Media Diagnosis and Treatment: Coherent Optical Detection of Middle Ear Disease
Brief Title: Coherent Optical Detection of Middle Ear Disease
Acronym: OCTII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other); National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Matthew Maksimoski, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 46057; 1R01DC019412-01A1 (NIH)
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Otitis Media; Otitis Media With Effusion; Otitis Media Acute
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Children's Wisconsin Urgent Care Clinics (Experimental): Subjects will receive a standard-of-care otoscopy examination, followed by a research-only examination using an OCT device (PCT).
  Interventions: Diagnostic Test: OCT Device(s)
- Children's Wisconsin (Effusion in 0 or 1 ear) (No Intervention): Subjects will only receive a standard-of-care otoscopy examination.
- Children's Wisconsin (Effusion in 2 ears) (Experimental): Subjects will receive standard-of-care ear and hearing examinations (otoscopy and audiometry/tympanometry), followed by research-only examinations using two OCT devices (UIUC OCT and PCT).
  Interventions: Diagnostic Test: OCT Device(s)

INTERVENTIONS:
Diagnostic Test: OCT Device(s) — Results from standard-of-care examinations will be compared to research-only examination(s) (OCT device(s)).
  Arms: Children's Wisconsin (Effusion in 2 ears); Children's Wisconsin Urgent Care Clinics

SUMMARY:
The purpose of this project is to see if optical coherence tomography (OCT), a new technology acting as an ultrasound for the ear, facilitates accurately diagnosing acute otitis media (AOM) and otitis media with effusion (OME) in children. Clinical diagnoses made using solely otoscopy will be compared to those made with the addition of OCT.

DETAILED DESCRIPTION:
Otitis media (OM) is the most common diagnosis in pediatric patients seen for illness in the United States, affects 90% of all children, and is the most common indication for antimicrobial therapy and surgery in young children. Despite many attempts to improve diagnosis, treatment, and prevention, OM continues its highly prevalent impact on children and substantial ongoing morbidity. OM continues as the most common cause of hearing loss in children and leads to speech, educational and other developmental delays. OM causes life-threatening complications and is expensive, resulting in over $5 billion annually in U.S. health care expenditures. Despite the prevalence and difficulties with OM, diagnostic accuracy to allow appropriate treatment is lacking, leading to misplaced resources in treating OM. This proposal builds on our central hypothesis that enhanced diagnostic tools, specifically, optical coherence tomography (OCT), will yield improved diagnosis and lead to reduced need for antibiotics to treat acute OM, reduced surgical interventions for chronic otitis media, and overall fewer complications and cost associated with this disease. In this proposal, the investigators will explore three specific aims. The first aim, part A, the investigators will perform a comparative assessment of middle ear pathology using otoscopy and OCT in pediatric patients that present to a primary care clinic with complaints of otalgia or OM, with the hypothesis that OCT added to standard otoscopy will improve diagnostic accuracy and reduce overall antibiotic prescriptions. In part B of this aim, a comparative assessment of middle ear pathology using otoscopy along with audiometry/tympanometry and OCT will be performed in pediatric patients that present to the pediatric otolaryngology clinic with a referral for chronic otitis media with effusion (OME), with the hypothesis that OCT added to standard otoscopy and audiometry/tympanometry will improve diagnostic accuracy and reduce overall need for surgery in patients with OME. In the second aim, using the OCT images captured in the previous aim, the investigators will develop image processing and machine learning algorithms for automated identification of effusions and biofilms in OCT image data to augment OM diagnosis for medical decision making. Finally, using the OCT images captured previously, along with our machine learning algorithms, the investigators will establish OCT B-mode and M-mode image-based features that predict the resolution or persistence of middle ear effusions over time. Collectively, this project will demonstrate how these advances in diagnostic tools and algorithms will improve diagnosis and provide added information for clinical decision making in the management of OM.

ELIGIBILITY:
Inclusion Criteria:

* Parental complaint of ear infection or ear pain (Children's Wisconsin Urgent Care Clinics) OR referred for evaluation of otitis media with effusion (Children's Wisconsin ENT Clinic)
* Speak English

Exclusion Criteria:

* Children with craniofacial abnormalities
* Children with diagnosed immunologic abnormalities
* Children with congenital syndromic conditions
* Current open and functioning ear tubes

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Children's Wisconsin Urgent Care Clinic Analysis (Standard-of-Care Diagnosis) | 5 years
  The investigators will look at the percentage of patients that receive the decision for antibiotic prescriptions using only a standard-of-care examination (otoscopy) (prior to addition of a research-only OCT device).
Children's Wisconsin Urgent Care Analysis (Research Device Diagnosis) | 5 years
  The investigators will look at the percentage of patients that receive the decision for antibiotic prescriptions after the addition of a research-only OCT device.
Children's Wisconsin ENT Clinic Analysis (Standard-of-Care Diagnosis) | 5 years
  The investigators will look at the percentage of patients that receive the decision for surgical intervention using only standard-of-care examinations (otoscopy, audiometry/tympanometry) (prior to addition of research-only OCT devices).
Children's Wisconsin ENT Clinic Analysis (Research Devices Diagnosis) | 5 years
  The investigators will look at the percentage of patients that receive the decision for surgical intervention after the addition of research-only OCT devices.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kerschner, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Children's Wisconsin ENT Clinic, Wauwatosa, Wisconsin
  - Children's Wisconsin Urgent Care Clinics, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerschner JE, Daley RA Jr, Link R, Jones RM, Peterson KJ, Chun RH, Flanary VA, Gorelik M, Keppel KL, Maksimoski M, Malloy M, Martin TJ, McCormick ME, Robey TC, Ansari S, Matoska GM, Rupcich CA, Saunderson ML, Shay SG, Sulman C, Erbe C, Thompson JK, Khampang P, Yan K, Simpson PM, Ho A, Monroy GL, Spillman DR, Aksamitiene E, Boppart SA. Clinical trial assessing the use of optical coherence tomography in decision making for children presenting with acute otitis media. Int J Pediatr Otorhinolaryngol. 2026 Jan 14;202:112728. doi: 10.1016/j.ijporl.2026.112728. Online ahead of print. PMID 41547297